CLINICAL TRIAL: NCT05487430
Title: The Effect of Self-Affirmation on Anxiety and Perceived Discomfort in Patients Who Underwent Open-Heart Surgery. A Randomized Controlled Trial
Brief Title: Self-Affirmation for Managing Anxiety and Perceived Discomfort in Open-Heart Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vic - Central University of Catalonia (Other)
Collaborators: Mehmet Akif Ersoy Thoracic and Cardiovascular Surgery and Research Hospital (Unknown); Trakya University (Other)
Responsible Party: Principal Investigator, Meltem Yildirim, Associated Professor, University of Vic - Central University of Catalonia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-52
Record Dates: First submitted 2022-07-21; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Surgery; Cardiac Disease
Keywords: anxiety; discomfort; open-heart surgery; self-affirmation; randomized controlled trial
MeSH Terms: conditions — Heart Diseases; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomised assignation of participants into two study groups: Intervention and Control.
Masking Description: Blinding the intervention group from the clinical staff and from the researchers was not possible due to the fact that the patients were listening to the affirmation recordings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Self-affirmation audio recording included 40 positive sentences in order to increase the sensation of well-being of the patients. Some examples are:
  1. Now I have decided to think more positively.
  2. I am in control of my thoughts.
  3. I am completely relaxed.
  4. I am strong, and I am aware of my strength.
  5. I can be comfortable and positive in any situation.
  6. I love myself as I am and accept myself for who I am.
  7. I know very well how to relax.
  8. All my muscles relax with every deep breath I take.
  9. I leave myself in peace.
  10. I am a relaxed, joyful, and happy person.
  11. I am calm at all times and in all situations.
  12. I know that everything that happens in my life happens for my own good.
  13. I am very good at relaxing.
  14. My life energy is rising.
  15. I am surrounded by positive energy.
  In the background of the recording there were sounds of birds crowing and river-like flowing water together for increasing the effect of relaxation.
  Interventions: Behavioral: Positive Self-Affirmation
- Control Group (No Intervention): The participants of the control group only received the conventional care given in the inpatient clinic.

INTERVENTIONS:
Behavioral: Positive Self-Affirmation — Each participant of the intervention group was given a set of earphones and an MP3 player which included an audio recording with a background sound of birds crowing and river-like flowing water together with the positive affirmation sentences. The self-affirmation sentences were created by the first author by paying special attention to not using negative predicates and words with negative meanings such as pain, nausea, and discomfort. In the audio recording, the affirmative sentences were verbalized by the first author with a soothing voice. Between each sentence, a pause is given so that the patient can repeat each sentence verbally or internally. The audio recording lasted 5 minutes 40 seconds and the patients were asked to listen to it at least once a day, however, they were encouraged to listen to it as much as they wanted.
  Arms: Intervention Group

SUMMARY:
This study adopted a randomized controlled pretest-posttest follow-up research design. The study was conducted at a public training and research hospital (Istanbul, Turkey) specialized in thoracic and cardiovascular surgery. The sample consisted of 61 patients randomized into two groups: intervention (n=34) and control (n=27). The participants of the intervention group listened to a self-affirmation audio recording for three days after surgery. Anxiety levels and perceived discomfort regarding pain, dyspnoea, palpitations, fatigue and nausea were measured daily. The study's main question is How do self-affirmation affect postoperative anxiety and perceived discomfort (regarding pain, dyspnoea, palpitations, fatigue and nausea) in patients who undergo open-heart surgery? In accordance with this question, the hypotheses was that repetitive positive self-affirmations decrease both anxiety and perceived discomfort in patients who underwent open-heart surgery.

DETAILED DESCRIPTION:
This study adopted a randomized controlled pretest-posttest follow-up research design in accordance with CONSORT guidelines with 2 study groups (intervention and control).

The study was conducted among the patients who underwent open-heart surgery in the in-patient clinics of a public hospital (Istanbul, Turkey). Following the surgical intervention, all patients were admitted to the cardiac intensive care unit (CICU) for close postoperative follow-up. According to the hospital protocol, the minimum duration for a CICU stay is 2 days after surgery in patients that are hemodynamically stabilized. On their 3rd postoperative day, they are discharged from CICU to be admitted to the in-patient clinic and; in this study, their first day in the clinic was considered as the adaptation and resting period, so that the sampling process was started on the 4th postoperative day.

Eighty-five patients were assessed for eligibility. Five patients excluded from the study before randomization. Following the randomization, 12 patients were excluded during the initial allocation and then 7 more patients were excluded during the follow-up. The final study sample consisted of 61 patients who underwent CABS; 34 in the intervention group and 27 in the control group.

The baseline data (pre-test) was obtained on the fourth postoperative day considering the fact that the patients were comfortably adapted to the in-patient clinic and were more open to collaborate in the study. Additionally, preoperative anxiety weren't considered as a baseline evaluation because it is known that during the preoperative period the sources of anxiety are mainly related to uncertainties and fear of death, however during the postoperative period the patients are more likely to be concerned about their need to be protected, in other words, their vulnerability and fragility.

Each patient was followed up for 3 days. The data collection process was lasted 4 months, between the 20th of November of 2019 and the 20th of March of 2020.

In this study, intention-to-treat analysis was not used as all the participants were asked to listen to the self-affirmation recording at least once a day, because daily repetition is the key element when affirming positive sentences in order to mobilize the inner sources of the individual. Therefore, only per-protocol analysis where all participants strictly adhered to the study protocol was conducted.

The data were analysed by using the Statistical Package for the Social Sciences (IBM, SPSS, 21.0) at a significance level of 0.05. In the descriptive analysis, mean was used for the numerical data, and frequency for the categorical data. The homogeneity between the study groups regarding the participants' descriptive characteristics was tested with the Chi-Square test. Repeated measures analysis of variance (ANOVA) was used to identify the differences between the study groups, meanwhile within-group comparisons were done by the Independent Sample t-Test. The power analyses conducted with G*Power indicated that this study had high power (1 - β = 0.93) with the effect size of d=0.91 (α=0,05).

ELIGIBILITY:
Inclusion Criteria:

* undergoing coronary artery bypass surgery for the first time,
* not having any history of a previous open cardiothoracic surgery
* being over 18 years
* being literate in Turkish.

Exclusion Criteria:

* having a diagnosed anxiety disorder
* having hearing deficiency
* having an emergency coronary artery bypass surgery
* staying in the cardiac intensive care unit for more than 48-hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Change in the level of state anxiety on 3 consecutive days | During 3 days, one measurement per day
  The primary outcome of the study was the level of state anxiety during the postoperative stay in the in-patient clinic. The State Trait Anxiety Inventory (STAI) was used to measure the level of anxiety. It is a 40 item, 4-point Likert scale ranging from 1 (not at all) to 4 (very much so) and consisting of two sub-dimensions; state anxiety and trait anxiety, 20 items each. The scale was developed by Spielberger et al. in 1970 and adapted to Turkish by Öner and LeCompte in 1983. The total score ranges from 20 to 80 where higher scores indicate higher levels of anxiety. For the subsequent measurements of anxiety, only the state dimension of the STAI was used.

SECONDARY OUTCOMES:
Change in the perceived level of pain on 3 consecutive days, measured by 0 to 10 numeric rating scale | During 3 days, one measurement per day
  Patients' level of perceived discomfort regarding pain was measured by a Numeric Rating Scale (NRS) of 0 to 10 where higher scores indicate more pain.
Change in the perceived level of dyspnoea on 3 consecutive days, measured by 0 to 10 numeric rating scale | During 3 days, one measurement per day
  Patients' level of perceived discomfort regarding dyspnoea was measured by a Numeric Rating Scale (NRS) of 0 to 10 where higher scores indicate more dyspnoea.
Change in the perceived level of palpitations on 3 consecutive days, measured by 0 to 10 numeric rating scale | During 3 days, one measurement per day
  Patients' level of perceived discomfort regarding palpitations was measured by a Numeric Rating Scale (NRS) of 0 to 10 where higher scores indicate more palpitations.
Change in the perceived level of fatigue on 3 consecutive days, measured by 0 to 10 numeric rating scale | During 3 days, one measurement per day
  Patients' level of perceived discomfort regarding fatigue was measured by a Numeric Rating Scale (NRS) of 0 to 10 where higher scores indicate more fatigue.
Change in the perceived level of nausea on 3 consecutive days, measured by 0 to 10 numeric rating scale | During 3 days, one measurement per day
  Patients' level of perceived discomfort regarding nausea was measured by a Numeric Rating Scale (NRS) of 0 to 10 where higher scores indicate more nausea.

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Yildirim, PhD, Principal Investigator — University of Vic - Central University of Catalonia
Locations (1):
- Mehmet Akif Ersoy Thoracic and Cardiovacular Surgery Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study will not be publicly available due to the privacy of the participants.

REFERENCES:
- [Background] Hernandez-Palazon J, Fuentes-Garcia D, Falcon-Arana L, Roca-Calvo MJ, Burguillos-Lopez S, Domenech-Asensi P, Jara-Rubio R. Assessment of Preoperative Anxiety in Cardiac Surgery Patients Lacking a History of Anxiety: Contributing Factors and Postoperative Morbidity. J Cardiothorac Vasc Anesth. 2018 Feb;32(1):236-244. doi: 10.1053/j.jvca.2017.04.044. Epub 2017 Apr 26. PMID 28803768
- [Background] Williams JB, Alexander KP, Morin JF, Langlois Y, Noiseux N, Perrault LP, Smolderen K, Arnold SV, Eisenberg MJ, Pilote L, Monette J, Bergman H, Smith PK, Afilalo J. Preoperative anxiety as a predictor of mortality and major morbidity in patients aged >70 years undergoing cardiac surgery. Am J Cardiol. 2013 Jan 1;111(1):137-42. doi: 10.1016/j.amjcard.2012.08.060. PMID 23245838
- [Background] Bang YY, Park H. Effects of auricular acupressure on the quality of sleep and anxiety in patients undergoing cardiac surgery: A single-blind, randomized controlled trial. Appl Nurs Res. 2020 Jun;53:151269. doi: 10.1016/j.apnr.2020.151269. Epub 2020 Apr 19. PMID 32451010
- [Background] Sherman DK. Self-Affirmation: Understanding the Effects. Soc Personal Psychol Compass 2013;7:834-45.
- [Background] Steele CM. The Psychology of Self-Affirmation: Sustaining the Integrity of the Self. 1988, 261-302.
- [Background] Sherman DK, Cohen GL. The Psychology of Self-defense: Self-Affirmation Theory. Advances in Experimental Social Psychology. 2006, 183-242.
- [Background] Creswell JD, Lam S, Stanton AL, Taylor SE, Bower JE, Sherman DK. Does self-affirmation, cognitive processing, or discovery of meaning explain cancer-related health benefits of expressive writing? Pers Soc Psychol Bull. 2007 Feb;33(2):238-50. doi: 10.1177/0146167206294412. PMID 17259584
- [Background] Yildirim M, Gulsoy H, Batmaz M, Ozgat C, Yesilbursali G, Aydin R, Ekiz S. Symptom Management: The Effects of Self-Affirmation on Chemotherapy-Related Symptoms. Clin J Oncol Nurs. 2017 Feb 1;21(1):E15-E22. doi: 10.1188/17.CJON.E15-E22. PMID 28107336
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c869. doi: 10.1136/bmj.c869. No abstract available. PMID 20332511
- [Background] Spielberger CD, Gorsuch RL, Lushene RE. Test Manual for the State Trait Anxiety Inventory. 1st Ed. California: Consulting Psychologists Press, 1970.
- [Background] Öner N, LeCompte AW. Stait Trait Anxiety Inventory Handbook (Süreksiz Durumluk/Sürekli Kaygı Envanteri El Kitabı). 1st Ed. Istanbul: Bogazici Universitesi Yayinlari, 1983.
- [Background] Gift AG, Narsavage G. Validity of the numeric rating scale as a measure of dyspnea. Am J Crit Care. 1998 May;7(3):200-4. PMID 9579246
- [Background] Gladman D, Nash P, Goto H, Birt JA, Lin CY, Orbai AM, Kvien TK. Fatigue numeric rating scale validity, discrimination and responder definition in patients with psoriatic arthritis. RMD Open. 2020 Jan;6(1):e000928. doi: 10.1136/rmdopen-2019-000928. PMID 31958274
- [Background] Wikstrom L, Nilsson M, Brostrom A, Eriksson K. Patients' self-reported nausea: Validation of the Numerical Rating Scale and of a daily summary of repeated Numerical Rating Scale scores. J Clin Nurs. 2019 Mar;28(5-6):959-968. doi: 10.1111/jocn.14705. Epub 2018 Nov 8. PMID 30357970
- [Background] Harden M, Nystrom B, Kulich K, Carlsson J, Bengtson A, Edvardsson N. Validity and reliability of a new, short symptom rating scale in patients with persistent atrial fibrillation. Health Qual Life Outcomes. 2009 Jul 15;7:65. doi: 10.1186/1477-7525-7-65. PMID 19604399
- [Background] Erturk EB, Unlu H. Effects of pre-operative individualized education on anxiety and pain severity in patients following open-heart surgery. Int J Health Sci (Qassim). 2018 Jul-Aug;12(4):26-34. PMID 30022900
- [Background] Robley L, Ballard N, Holtzman D, Cooper W. The experience of stress for open heart surgery patients and their caregivers. West J Nurs Res. 2010 Oct;32(6):794-813. doi: 10.1177/0193945910361469. Epub 2010 Aug 9. PMID 20696847
- [Background] Feuchtinger J, Burbaum C, Heilmann C, Imbery C, Siepe M, Stotz U, Fritzsche K, Beyersdorf F. Anxiety and fear in patients with short waiting times before coronary artery bypass surgery--a qualitative study. J Clin Nurs. 2014 Jul;23(13-14):1900-7. doi: 10.1111/jocn.12467. Epub 2013 Dec 27. PMID 24372741
- [Background] Karlsson AK, Mattsson B, Johansson M, Lidell E. Well-being in patients and relatives after open-heart surgery from the perspective of health care professionals. J Clin Nurs. 2010 Mar;19(5-6):840-6. doi: 10.1111/j.1365-2702.2009.03017.x. PMID 20500327
- [Background] Karlsson AK, Johansson M, Lidell E. Fragility--the price of renewed life. Patients experiences of open heart surgery. Eur J Cardiovasc Nurs. 2005 Dec;4(4):290-7. doi: 10.1016/j.ejcnurse.2005.03.009. PMID 15886056
- [Background] Lapum J, Angus JE, Peter E, Watt-Watson J. Patients' discharge experiences: returning home after open-heart surgery. Heart Lung. 2011 May-Jun;40(3):226-35. doi: 10.1016/j.hrtlng.2010.01.001. Epub 2010 Apr 14. PMID 20561868
- [Background] Leon C. Raise Your Energy for Mind Body Wellness Chakra Biokinetics. Morrisville: Lulu, 2006, 81-2.
- [Background] Chandler CK, Holden JM, Kolander CA. Counseling for Spiritual Wellness: Theory and Practice. J Couns Dev 1992;71:168-75.
- [Background] Tripepi G, Chesnaye NC, Dekker FW, Zoccali C, Jager KJ. Intention to treat and per protocol analysis in clinical trials. Nephrology (Carlton). 2020 Jul;25(7):513-517. doi: 10.1111/nep.13709. Epub 2020 Mar 15. PMID 32147926
- [Background] World Medical Association.. World Medical Association Declaration of Helsinki. Ethical principles for medical research involving human subjects. Bull World Health Organ. 2001;79(4):373-4. Epub 2003 Jul 2. No abstract available. PMID 11357217
- [Background] Tully PJ, Bennetts JS, Baker RA, McGavigan AD, Turnbull DA, Winefield HR. Anxiety, depression, and stress as risk factors for atrial fibrillation after cardiac surgery. Heart Lung. 2011 Jan-Feb;40(1):4-11. doi: 10.1016/j.hrtlng.2009.12.010. Epub 2010 May 8. PMID 20561864
- [Background] Miozzo AP, Stein C, Bozzetto CB et al. Massage therapy reduces pain and anxiety after cardiac surgery: A systematic review and meta-analysis of randomized clinical trials. Clin Trials Regul Sci Cardiol 2016;23-24:1-8.
- [Background] Aygin D, Sen S. Acupressure on Anxiety and Sleep Quality After Cardiac Surgery: A Randomized Controlled Trial. J Perianesth Nurs. 2019 Dec;34(6):1222-1231. doi: 10.1016/j.jopan.2019.03.014. Epub 2019 Jul 11. PMID 31303389
- [Background] Voss JA, Good M, Yates B, Baun MM, Thompson A, Hertzog M. Sedative music reduces anxiety and pain during chair rest after open-heart surgery. Pain. 2004 Nov;112(1-2):197-203. doi: 10.1016/j.pain.2004.08.020. PMID 15494201
- [Background] Heidari S, Babaii A, Abbasinia M, Shamali M, Abbasi M, Rezaei M. The Effect of Music on Anxiety and Cardiovascular Indices in Patients Undergoing Coronary Artery Bypass Graft: A Randomized Controlled Trial. Nurs Midwifery Stud. 2015 Dec;4(4):e31157. doi: 10.17795/nmsjournal31157. Epub 2015 Dec 1. PMID 26835471
- [Background] İbrahimoğlu Ö, Kanan N. The Effect of Progressive Muscle Relaxation Exercises After Endotracheal Extubation on Vital Signs and Anxiety Level in Open Heart Surgery Patients. Turkish J Intensive Care 2017;15:98-106.
- [Background] Shifeng L, Yiling W, Fumin Z et al. Self-affirmation buffering by the general public reduces anxiety levels during the COVID-19 epidemic. Acta Psychol Sin 2020;52:886.
- [Background] Sherman DK, Bunyan DP, Creswell JD, Jaremka LM. Psychological vulnerability and stress: the effects of self-affirmation on sympathetic nervous system responses to naturalistic stressors. Health Psychol. 2009 Sep;28(5):554-62. doi: 10.1037/a0014663. PMID 19751081
- [Background] Morgan JI, Harris PR. Evidence that brief self-affirming implementation intentions can reduce work-related anxiety in downsize survivors. Anxiety Stress Coping. 2015;28(5):563-75. doi: 10.1080/10615806.2015.1004665. Epub 2015 Feb 4. PMID 25575334
- [Background] Harris PR, Mayle K, Mabbott L, Napper L. Self-affirmation reduces smokers' defensiveness to graphic on-pack cigarette warning labels. Health Psychol. 2007 Jul;26(4):437-46. doi: 10.1037/0278-6133.26.4.437. PMID 17605563
- [Background] Chen WJ, Nelson AM, Johnson HB, Fleming R. Effects of self-affirmation on emotion and cardiovascular responses. Stress Health. 2021 Apr;37(2):201-212. doi: 10.1002/smi.2986. Epub 2020 Sep 24. PMID 32954655
- [Background] Huang AP, Sakata RK. Pain after sternotomy - review. Braz J Anesthesiol. 2016 Jul-Aug;66(4):395-401. doi: 10.1016/j.bjane.2014.09.013. Epub 2016 Apr 23. PMID 27343790
- [Background] Broderick JE, Junghaenel DU, Schwartz JE. Written emotional expression produces health benefits in fibromyalgia patients. Psychosom Med. 2005 Mar-Apr;67(2):326-34. doi: 10.1097/01.psy.0000156933.04566.bd. PMID 15784801
- [Background] Norman SA, Lumley MA, Dooley JA, Diamond MP. For whom does it work? Moderators of the effects of written emotional disclosure in a randomized trial among women with chronic pelvic pain. Psychosom Med. 2004 Mar-Apr;66(2):174-83. doi: 10.1097/01.psy.0000116979.77753.74. PMID 15039501
- [Background] Bauer BA, Cutshall SA, Anderson PG, Prinsen SK, Wentworth LJ, Olney TJ, Messner PK, Brekke KM, Li Z, Sundt TM 3rd, Kelly RF, Bauer BA. Effect of the combination of music and nature sounds on pain and anxiety in cardiac surgical patients: a randomized study. Altern Ther Health Med. 2011 Jul-Aug;17(4):16-23. PMID 22314630
- [Background] Johnson D, Hurst T, Thomson D, Mycyk T, Burbridge B, To T, Mayers I. Respiratory function after cardiac surgery. J Cardiothorac Vasc Anesth. 1996 Aug;10(5):571-7. doi: 10.1016/s1053-0770(96)80130-3. PMID 8841860
- [Background] Neuman A, Gunnbjornsdottir M, Tunsater A, Nystrom L, Franklin KA, Norrman E, Janson C. Dyspnea in relation to symptoms of anxiety and depression: A prospective population study. Respir Med. 2006 Oct;100(10):1843-9. doi: 10.1016/j.rmed.2006.01.016. Epub 2006 Mar 3. PMID 16516455
- [Background] Nikolajsen L, Jensen TS. Phantom limb pain. Br J Anaesth. 2001 Jul;87(1):107-16. doi: 10.1093/bja/87.1.107. No abstract available. PMID 11460799
- [Background] Tang D, Schmeichel BJ. Self-affirmation facilitates cardiovascular recovery following interpersonal evaluation. Biol Psychol. 2015 Jan;104:108-15. doi: 10.1016/j.biopsycho.2014.11.011. Epub 2014 Dec 8. PMID 25498787
- [Background] Ai AL, Wink P, Shearer M. Fatigue of survivors following cardiac surgery: positive influences of preoperative prayer coping. Br J Health Psychol. 2012 Nov;17(4):724-42. doi: 10.1111/j.2044-8287.2012.02068.x. Epub 2012 Apr 23. PMID 22524258
- [Background] Sawatzky JA, Rivet M, Ariano RE, Hiebert B, Arora RC. Post-operative nausea and vomiting in the cardiac surgery population: who is at risk? Heart Lung. 2014 Nov-Dec;43(6):550-4. doi: 10.1016/j.hrtlng.2014.07.002. Epub 2014 Aug 21. PMID 25151430
- [Background] Lavi R, Katznelson R, Cheng D, Minkovich L, Klein A, Carroll J, Karski J, Djaiani G. The effect of nasogastric tube application during cardiac surgery on postoperative nausea and vomiting--a randomized trial. J Cardiothorac Vasc Anesth. 2011 Feb;25(1):105-9. doi: 10.1053/j.jvca.2010.02.011. Epub 2010 Apr 27. PMID 20427207
- [Background] Mace L. An audit of post-operative nausea and vomiting, following cardiac surgery: scope of the problem. Nurs Crit Care. 2003 Sep-Oct;8(5):187-96. doi: 10.1046/j.1362-1017.2003.00029.x. PMID 14653525
- [Background] Rodrigues HF, Furuya RK, Dantas RAS, Rodrigues AJ, Dessotte CAM. Association of preoperative anxiety and depression symptoms with postoperative complications of cardiac surgeries. Rev Lat Am Enfermagem. 2018 Nov 29;26:e3107. doi: 10.1590/1518-8345.2784.3107. PMID 30517589
- [Background] Unverzagt S, Prondzinsky R, Peinemann F. Single-center trials tend to provide larger treatment effects than multicenter trials: a systematic review. J Clin Epidemiol. 2013 Nov;66(11):1271-80. doi: 10.1016/j.jclinepi.2013.05.016. Epub 2013 Aug 20. PMID 23972520
- [Background] Forgeard MJC, Seligman MEP. Seeing the glass half full: A review of the causes and consequences of optimism. Prat Psychol 2012;18:107-20.
- [Derived] Yildirim M, Akbal S, Turkoglu M. The effect of self-affirmation on anxiety and perceived discomfort in patients who have undergone open-heart surgery. A randomized controlled trial. Appl Nurs Res. 2023 Aug;72:151687. doi: 10.1016/j.apnr.2023.151687. Epub 2023 May 17. PMID 37423676